CLINICAL TRIAL: NCT05628935
Title: The Effect of Anesthesia Method on Neutrophil-Lymphocyte Ratio in Patients Undergoing Forearm Surgery
Brief Title: Effect of Anesthesia Method on Neutrophil-Lymphocyte Ratio
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Bengü Gülhan Köksal, medical doctor, Zonguldak Bulent Ecevit University
Other Study IDs: 2020-22/17
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Inflammation; Anesthesia
Keywords: General Anesthesia; Neutrophil Lymphocyte Ratio; Peripheral Nerve Block
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group G: Patients Undergoing Forearm Surgery under general anesthesia
- Group P: Patients Undergoing Forearm Surgery under peripheral nerve block
  Interventions: Procedure: peripheral nerve block

INTERVENTIONS:
Procedure: peripheral nerve block — local anesthetic application to the brachial plexus
  Groups: Group P

SUMMARY:
The neutrophil/lymphocyte ratio (NLR) is a simple and inexpensive marker of the inflammatory response. NLR is affected not only by surgical trauma but also by the anesthetic method. The method of anesthesia can affect NLR, thereby modulating the inflammatory response and surgical outcomes. In this study, it was aimed to evaluate the relationship between blood NLR and anesthesia techniques in patients undergoing forearm surgery, and the secondary aim was to evaluate the relationship between Platelet/lymphocyte ratio (TLR), Mean Platelet Volume (MPV) and anesthesia techniques.

ELIGIBILITY:
Inclusion Criteria:

* Underwent forearm surgery
* Between aged 18-70
* Under general anesthesia or peripheral nerve block

Exclusion Criteria:

* acute infection
* morbid obesity
* chronic treatment with steroids or immunosuppressants
* recently received chemotherapy
* hepatic and renal dysfunction;
* chronic alcohol abusers
* Multiple trauma
* Patients with missing data in their files

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-65 years who have underwent forearm surgery
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Neutrophil/lymphocyte ratio | up to 24 hours after surgery
  Differences in neutrophil-lymphocyte ratio between patients who underwent general anesthesia and peripheral nerve block

SECONDARY OUTCOMES:
Platelet/lymphocyte ratio | up to 24 hours after surgery
  Differences in Platelet/lymphocyte ratio between patients who underwent general anesthesia and peripheral nerve block
Mean Platelet Volume | up to 24 hours after surgery
  Differences in Mean Platelet Volume between patients who underwent general anesthesia and peripheral nerve block

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University Medicine Faculty, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No